CLINICAL TRIAL: NCT06599762
Title: Evaluation of Tranexamic Acid Among Outpatients With Myelodysplastic Syndromes and Acute Myeloid Leukemia: a Multicenter Pilot Trial
Brief Title: Evaluation of Tranexamic Acid in Myelodysplastic Syndromes and Acute Myeloid Leukemia
Acronym: MYELO-CAN:TXA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Brett Houston, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHI-001-1
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
Keywords: Tranexamic Acid; Randomized Controlled Trial; Myelodysplastic Syndrome; Acute Myeloid Leukemia; Thrombocytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Thrombocytopenia | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid (Experimental)
  Interventions: Drug: Tranexamic acid
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid 1000mg orally two or three times daily
  Arms: Tranexamic Acid
Drug: Placebo — Placebo orally two or three times daily
  Arms: Matching Placebo

SUMMARY:
Myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML) are serious, life changing blood cancers. Patients with MDS and AML commonly experience complications related to bleeding, which affect patient quality-of-life and can sometimes lead to hospitalization or death. The investigators will conduct a randomized controlled trial to evaluate the effectiveness and safety of tranexamic acid (TXA; a medication that prevents clots from dissolving) to prevent bleeding. In this study, 50% of patients will be randomized (like the flip of a coin) to receive TXA; the other 50% of patients will receive placebo. The investigators will monitor both groups of patients to see if the medication improves the risk and/or severity of bleeding. If tranexamic acid were to safely reduced the frequency of bleeding, this would broadly influence how doctors provide care for patients with MDS and AML around the world.

DETAILED DESCRIPTION:
RATIONALE: Myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML) are serious, life-changing blood cancers. Despite the best efforts of their care team, patients with MDS and AML commonly experience complications related to bleeding. These complications affect patient quality-of-life and can sometimes lead to hospitalization or death. Evaluation of affordable and widely available treatments to minimize bleeding complications among patients with MDS and AML is needed.

STUDY OBJECTIVES: To evaluate the feasibility of tranexamic acid (TXA) that will evaluate the efficacy and safety of treatments to minimize bleeding in patients with MDS and AML treated in the outpatient setting.

METHODOLOGY: The investigators will conduct a multicenter pilot randomized control trial (RCT) for outpatients ≥18 years of age with MDS and AML. Patients with MDS and AML with low platelet counts will receive TXA (a medication that prevents clots from dissolving). TXA is commonly used in other clinical settings but have not been studied in patients with MDS or AML receiving outpatient chemotherapy (ie, chemotherapy that can be given from clinic, rather than a hospital). In this study, 50% of patients will be randomized (like the flip of a coin) to receive the medication the investigators are studying. The other 50% of patients will receive a matching placebo.

OUTCOMES: The primary feasibility outcome is the ability to enroll a mean of 1 patient per site per month.

SITES AND DURATION: The investigators will initially enroll patients from 10-15 sites across Canada. The expected duration of enrollment is 2 years.

SIGNIFICANCE: With a broad range of stakeholders, including patient partners, the trial will address a broadly applicable patient-prioritized question. Tranexamic acid is readily available, inexpensive, and has an established side effect profile. Results of this trial are highly generalizable and will broadly impact the care of patients with MDS and AML.

ELIGIBILITY:
Inclusion Criteria:

Master platform inclusion criteria:

1. Age ≥ 18 years
2. Diagnosis of myelodysplastic syndromes or acute myeloid leukemia

MYELO-CAN TXA inclusion criteria:

1. Receipt of less-intensive chemotherapy (includes both frontline and relapsed/refractory setting)
2. Severe thrombocytopenia (platelets ≤ 30x10^9/L or platelets ≤ 50x10^9/L prior to chemotherapy initiation)

Exclusion Criteria:

Master platform exclusion criteria:

1. Participant is deemed unlikely to survive >30 days (as determined by clinical team)
2. Participant unable to provide informed consent

MYELO-CAN TXA exclusion criteria:

1. Known allergy to tranexamic acid
2. Active thromboembolic disease
3. Active ischemic heart disease
4. Gross hematuria
5. Stage V chronic kidney disease
6. Clinically suspected disseminated intravascular coagulation (DIC)
7. Pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient enrollment feasibility | 2 months
  The ability to enroll a median of 1 patient per site per month (10 patients / month when all sites are active)

SECONDARY OUTCOMES:
Venous or arterial thromboembolism incidence | 2 months
  The incidence of venous or arterial thromboembolism will be measured as a safety outcome.
Catheter-associated thrombosis incidence | 2 months
  The incidence of catheter-associated thrombosis will be measured as a safety outcome.
Study drug discontinuation | 2 months
  Study drug discontinuation due to adverse events will be measured as a safety outcome.
Ability to consent 30% of eligible patients | 2 months
  The ability to consent 30% of eligible patients will be measured as a feasibility outcome.
Grade 3 and 4 nausea/vomiting | 2 months
  The incidence of grade 3 and 4 nausea/vomiting (CTCAE) will be measured as a safety outcome.
Visual disturbance incidence | 2 months
  The incidence of new visual disturbances will be measured as a safety outcome.
Medication adherence | 2 months
  Protocol adherence of 80% of all intended medication doses per patient will be measured as a feasibility outcome.

OTHER OUTCOMES:
Quality of life evaluation using PROMIS questionnaire | 2 months
  Quality of life evaluation at baseline and monthly using the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue SF7a patient questionnaire.
Quality of life evaluation using EORTC questionnaire | 2 months
  Quality of life evaluation at baseline and monthly using the Core Quality of Life Questionnaire of the European Organisation For Research And Treatment Of Cancer (EORTC) C30 questionnaire.
Grade 2 to 5 bleeding incidence | 2 months
  The incidence of World Health Organization (WHO) defined grade 2 to 5 bleeding will be measured as a tertiary clinical outcome.
WHO bleeding incidence | 2 months
  The incidence of World Health Organization (WHO) bleeding stratified by grade will be measured as a clinical outcome.
Red blood cell transfusion exposure | 2 months
  The proportion of patients transfused red blood cells (RBC) will be measured as a clinical outcome.
Red blood cell transfusion volume | 2 months
  The mean/median number of red blood cell units transfused per patient will be measured as a clinical outcome.
Platelet transfusion volume | 2 months
  The mean/median number of platelet doses administered per patient will be measured as a clinical outcome.
Platelet transfusion exposure | 2 months
  The proportion of patients transfused with platelets will be measured as a clinical outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada